CLINICAL TRIAL: NCT03607344
Title: Day-case Laparoscopic Sacrocolpopexy, a Compelling Option in Selected Patients
Brief Title: Day Case Laparoscopic Sacrocolpopexy, a New Management
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: URO-BASE04
Record Dates: First submitted 2018-07-23; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: Sacrocolpopexy; Day case surgery; Laparoscopic
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Cohort — Patients undergoing ambulatory laparoscopic sacrocolpopexy

SUMMARY:
Facing the stakes of hospital beds, this study assessed day case variant technic of laparoscopic sacrocolpopexy with or without robotic assistant.

DETAILED DESCRIPTION:
Pelvic organ prolapse (POP) is an increasingly common functional disorder which affects approximately 40% of female population. Of these 12% are symptomatic and suffer of physical and emotional distress. 11% will undergo a surgical procedure. Since its introduction by Lane in 1982, Sacrocolpopexy (SCP) became the surgical "gold standard" for correcting vaginal vault .

With minimal invasive approach, SCP had an mean hospitalization time of 3 to 7 days .

With rising health care cost and its inherent economic burden, safe and viable options to reduce cost must be sought.

Day case surgery has developed rapidly in the USA since the 1970s, and has spread to Europe, especially in Great Britain. But the High Authority of Health in France found a delay in its development.

In view of the evolution of surgical and anesthetic techniques, and the low complication rate of SCP, it seemed natural to imagine that this intervention could be done in an ambulatory setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic anterior, apical and/or posterior compartment prolapse
* Patients with stage 2 or greater, according to the POP-Q classification
* Patients with a body mass index (BMI) < 30
* Patients with an American Society of Anesthesiologist (ASA) score < ou = 3.

Exclusion Criteria:

* Patient with prior history of pelvic cancer surgery and radiotherapy of the pelvis

Ages: 30 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort is selected from the investigators institution. All consecutive patients undergoing ambulatory laparoscopic sacrocolpopexy performed by two experimented urologist surgeons at the investigators university hospital, with an ambulatory department, was enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-01-26 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The success rate of outpatient laparoscopic sacrocolpopexy | 1 month post-operative
  The success rate of outpatient sacrocolpopexy is defined by the number of patients who leaves hospital at the day of surgery

SECONDARY OUTCOMES:
Post-operative adverses events | 1 month post-operative
  Adverses events are readmission, hospitalization at another medical hospitalization, complication and if patient has consulted her primary care practitioner or in the emergency department